CLINICAL TRIAL: NCT07020299
Title: Effect of Trans-cutenuous Electrical Diaphragmatic Stimulation on Severe Chronic Obstructive Pulmonary Disease Exacerbation
Brief Title: Effect of Electrical Diaphragmatic Stimulation on Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine department faculty of medicine mansoura university, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD.24.08.878
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diaphragm Electrical Activity; COPD (Chronic Obstructive Pulmonary Disease)
Keywords: chronic obstructive pulmonary disease exacerbation; Electrical diaphragmatic stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Effect of trans-cutenuous electrical diaphragmatic stimulation on severe chronic obstructive pulmonary disease exacerbation
Who Masked: Care Provider
Masking Description: Participants will be randomly assigned into a TEDS group or control group. Method of randomization : Before participant recruitment, sequential sealed envelopes are prepared by an independent investigator, with one envelope will be chosen randomly by another investigator for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEDS group will be subjected to sessions of TEDS (Active Comparator): TEDS group will be subjected to sessions of TEDS as follow : Digital electrical muscle stimulator (EV-906 Digital TENS/EMS made in TAIWAN) is applied to induce diaphragm contraction.
  Interventions: Device: Device : Digital electrical muscle stimulator is applied to induce diaphragm contraction.
- Non TEDS group will not be subjected to sessions of TEDS (No Intervention): Non TEDS group will not be subjected to sessions of TEDS

INTERVENTIONS:
Device: Device : Digital electrical muscle stimulator is applied to induce diaphragm contraction. — TEDS group will be subjected to sessions of TEDS as follow : Digital electrical muscle stimulator (EV-906 Digital TENS/EMS made in TAIWAN) is applied to induce diaphragm contraction.
  Arms: TEDS group will be subjected to sessions of TEDS

SUMMARY:
Respiratory muscle dysfunction is a common consequence of chronic obstructive pulmonary disease (COPD).

This technique consists of placing electrodes on the skin at locations near the motor points of the diaphragm, transmitting an intermittent current, and generating action potentials capable of producing muscle contractions

DETAILED DESCRIPTION:
Respiratory muscle dysfunction is a common consequence of chronic obstructive pulmonary disease (COPD).Weakness or fatigue of the diaphragm and accessory muscles of inspiration is widely recognized in patients on mechanical ventilation. There is increasing evidence to show mechanical ventilation itself may adversely affect the diaphragm's structure and function, which has been termed ventilator-induced diaphragmatic dysfunction. However, in patients with more severe COPD, the benefits of rehabilitation may be limited. In this context, there are new approaches to PR, such as electrical stimulation, a technique that externally stimulates contractions of peripheral muscles to improve peripheral muscle function in patients with severe COPD. This technique consists of placing electrodes on the skin at locations near the motor points of the diaphragm, transmitting an intermittent current, and generating action potentials capable of producing muscle contractions

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Known cases of COPD admitted at respiratory critical care unit with severe acute exacerbation (defined according to GOLD 2024).

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m2
* Post arrest patients
* Brain death
* Hemodynamic instability
* Invasive MV
* Lung disease other than COPD
* Pregnancy , ascitis.
* History of neuromuscular disease at admission
* Spinal injuries
* Skin lesions or an open lesion in the regions where the electrodes would be placed
* Use of pacemakers
* Patients on maintenance steroid therapy
* Depletating disease as malignancy 14. Patients refusing the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the progression to invasive mechanical ventilation(IMV) | 6 months
  Functional assessment by US measurement of diaphragmatic excursion and thickness fraction in (cm) including base line measurement and post treatment measurement ( at the end of admission).

SECONDARY OUTCOMES:
The secondary outcomes is the duration of ICU admission | 12 months
  The secondary outcomes is the duration of ICU admission (days), the immediate effect of TEDS and after sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, lecturer, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Faculty of medicine mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No